CLINICAL TRIAL: NCT07012577
Title: Observational Study on the Accuracy and Completeness of General Artificial Intelligence in the Diagnosis and Therapeutic Recommendations for Failed or Painful Total Hip Arthroplasty
Brief Title: Observational Study on AI Accuracy in Diagnosing and Treating Failed or Painful Hip Arthroplasty
Acronym: PAINGPT
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, francesco castagnini, Principal investigator, Istituto Ortopedico Rizzoli
Other Study IDs: 203/2025/Oss/IOR
Record Dates: First submitted 2025-05-31; First posted 2025-06-10 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Total Hip Arthroplasty (THA)
Keywords: Artificial intelligence; total hip arthroplasty; diagnosis; treatment
MeSH Terms: conditions — Disease | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Failed or Painful Total Hip Arthroplasty Patients: Patients with documented failed/painful THA (aseptic loosening, infection, fracture, etc.) selected from a tertiary center database (2004-2024).
  Interventions: Other: GPT-4 Assessment; Other: Arthroplasty Fellow Assessment; Other: Specializing Resident (4th year) Assessment; Other: Junior Resident (3rd year) Assessment

INTERVENTIONS:
Other: GPT-4 Assessment — Diagnostic/Prognostic evaluation of any single case provided by AI (GPT-4). GPT-4 provides diagnosis/treatment recommendations via standardized prompts
Other: Arthroplasty Fellow Assessment — Diagnostic/Prognostic evaluation of any single case provided by an human expert
Other: Specializing Resident (4th year) Assessment — Diagnostic/Prognostic evaluation of any single case provided by an human expert
Other: Junior Resident (3rd year) Assessment — Diagnostic/Prognostic evaluation of any single case provided by an human expert

SUMMARY:
Primary Goal:

This study aims to evaluate the diagnostic and therapeutic accuracy of GPT-4 (an advanced AI language model) compared to three orthopedic surgeons with varying experience levels in cases of failed or painful total hip arthroplasty.

Key Research Questions:

Diagnostic Accuracy:

Does GPT-4 provide correct, partially correct, or incorrect diagnoses compared to human orthopaedic surgeons?

Diagnostic Completeness:

Are GPT-4's diagnostic suggestions complete, partially complete, or incomplete compared to those of orthopedic surgeons?

Treatment Accuracy:

Does GPT-4 recommend correct, partially correct, or incorrect treatments for failed hip arthroplasty?

Treatment Completeness:

Are GPT-4's treatment recommendations fully comprehensive, partially complete, or incomplete compared to those of orthopaedic surgeon?

Study Design:

Participants:

20 anonymized patient cases (ages 18-80) with failed or painful hip arthroplasties, treated at IRCCS Istituto Ortopedico Rizzoli (Bologna, Italy) between 2004-2024.

Cases were selected based on clear diagnostic and treatment records (no ambiguous or incomplete data).

Comparison Groups:

GPT-4 (via ChatGPT interface)

Three orthopedic doctors (with different experience levels: resident, specialist, senior surgeon)

Method:

Each case (clinical summary + X-ray image) is presented to GPT-4 and the three doctors.

They must provide a diagnosis and treatment recommendations.

Two independent evaluators (principal investigator + department head) blindly assess responses for correctness and completeness using a 3-point scale (0=wrong/incomplete, 2=correct/complete).

Statistical analysis compares GPT-4 vs. human performance.

Expected Outcomes:

Determine if AI can match or outperform doctors in diagnosing and treating hip arthroplasty failures.

Assess whether GPT-4 could serve as a supplementary tool in orthopedic decision-making.

Ethical & Privacy Considerations:

No real-time patient data is used-only anonymized past cases.

No personal/sensitive data is shared with OpenAI (GPT-4 is used via a standard web interface).

Study complies with GDPR, HIPAA, and ethical AI guidelines.

Timeline:

Study duration: ~8 months (from ethics approval to final analysis).

Results will be published regardless of outcome.

Why This Study Matters:

First study evaluating GPT-4's role in complex orthopedic diagnostics.

Could influence future AI-assisted clinical decision-making in joint replacement surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 and ≤80 years old).
* Documented painful or failed total hip arthroplasty requiring clinical/radiological evaluation (2004-2024).
* Complete pre-operative clinical history, imaging (X-ray/tomography), and surgical reports.
* Clear diagnosis of failure mode (e.g., aseptic loosening, infection, fracture, wear).
* Treatment and outcomes fully documented in the institutional database.
* "Exemplary" cases with minimal diagnostic ambiguity (per Engh/MusculoSkleletal Infection Society criteria, etc.).

Exclusion Criteria:

* total hip arthroplasty with no documented failure/pain (well-functioning implants).
* Incomplete clinical/radiological records (e.g., missing pre-operative imaging or surgical notes).
* Complex/multifactorial failures (e.g., concurrent infection + loosening + fracture).
* Radiographs/images non-interpretable (poor quality, missing views).
* Cases with conflicting diagnoses/treatments in original records.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study evaluated 20 anonymized cases of failed/painful total hip arthroplasty (2004-2024) from a tertiary center. Cases were selected for diagnostic clarity (e.g., aseptic loosening, periprosthetic fracture) and excluded if records were incomplete or ambiguous. Two senior surgeons verified case eligibility. Each case was assessed by GPT-4, an arthroplasty fellow, a 4th-year resident, and a 3rd-year resident for diagnostic/therapeutic accuracy.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic correctness | Immediate (post-case evaluation)
  Proportion of fully correct diagnoses (score=2) by each rater, Scale 0 (worst outcome) - 2 (best outcome). 0: incorrect, 1: imprecise, 2: correct
Diagnostic completeness | Immediate (post-case evaluation)
  Proportion of fully complete diagnoses (score=2). Scale 0 (worst outcome) - 2 (best outcome). 0: incomplete, 1: partially complete, 2: complete
Treatment recommendation correctness | Immediate (post-case evaluation)
  Proportion of fully correct treatments (score=2) by each rater. Scale 0 (worst outcome) - 2 (best outcome). 0: incorrect, 1: imprecise, 2: correct
Treatmetn recommendation completeness | Immediate (post-case evaluation)
  Proportion of fully complete treatments (score=2). Scale 0 (worst outcome) - 2 (best outcome). 0: incomplete, 1: partially complete, 2: complete

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Castagnini, MD, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- SC Ortopedia e Traumatologia e Chirurgia Protesica e dei Reimpianti di Anca e Ginocchio, IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Rater evaluations on clinical cases; no direct patient data are included; all datasets are anonymized and do not allow identification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Immediately upon publication. Access limit: indefinitely
Access Criteria: With researchers, clinicians, or institutions upon request or directly via public repository.
URL: https://doi.org/10.5281/zenodo.15564513

REFERENCES:
- [Background] Knee CJ, Campbell RJ, Graham DJ, Handford C, Symes M, Sivakumar BS. Examining the role of ChatGPT in the management of distal radius fractures: insights into its accuracy and consistency. ANZ J Surg. 2024 Jul-Aug;94(7-8):1391-1396. doi: 10.1111/ans.19143. Epub 2024 Jul 5. PMID 38967407
- [Background] Dagher T, Dwyer EP, Baker HP, Kalidoss S, Strelzow JA. "Dr. AI Will See You Now": How Do ChatGPT-4 Treatment Recommendations Align With Orthopaedic Clinical Practice Guidelines? Clin Orthop Relat Res. 2024 Dec 1;482(12):2098-2106. doi: 10.1097/CORR.0000000000003234. Epub 2024 Sep 6. PMID 39246048
- [Background] Artioli E, Veronesi F, Mazzotti A, Brogini S, Zielli SO, Giavaresi G, Faldini C. Assessing ChatGPT responses to common patient questions regarding total ankle arthroplasty. J Exp Orthop. 2024 Dec 31;12(1):e70138. doi: 10.1002/jeo2.70138. eCollection 2025 Jan. PMID 39741912
- [Background] Pagano S, Strumolo L, Michalk K, Schiegl J, Pulido LC, Reinhard J, Maderbacher G, Renkawitz T, Schuster M. Evaluating ChatGPT, Gemini and other Large Language Models (LLMs) in orthopaedic diagnostics: A prospective clinical study. Comput Struct Biotechnol J. 2024 Dec 26;28:9-15. doi: 10.1016/j.csbj.2024.12.013. eCollection 2025. PMID 39850460

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT07012577/Prot_SAP_000.pdf